CLINICAL TRIAL: NCT06691594
Title: Prospective, Single-arm, Phase II Study of Stereotactic Radiotherapy Combined with PD-1 Monoclonal Antibody and Chemotherapy As Neoadjuvant Treatment for Triple-negative Breast Cancer
Brief Title: Neoadjuvant Treatment of Triple-Negative Breast Cancer with Stereotactic Radiotherapy, PD-1 Monoclonal Antibody, and Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4456
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Invasive
Keywords: preoperative radiothrapy; immunotherapy; triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant SBRT combined with PD-1 monoclonal antibody and chemotherapy (Experimental): Eligible participants will receive neoadjuvant treatment consisting of:
  SBRT: One session of 10Gy radiation to the primary tumor, followed by a 150mg subcutaneous injection of pembrolizumab (PD-1 inhibitor).
  Chemotherapy and Immunotherapy: One week after SBRT, participants will undergo 6 cycles of pembrolizumab (400mg), albumin-bound paclitaxel (250mg/m²), and carboplatin (AUC=5).
  Surgery: Surgery will be performed 21 days after the last chemotherapy cycle, with either breast-conserving surgery or modified radical mastectomy. Pathological evaluation will assess the treatment response.
  Adjuvant Immunotherapy: Four weeks post-surgery, patients will receive pembrolizumab every 3 weeks for up to 1 year.
  Interventions: Radiation: neoadjuvant SBRT combined with PD-1 monoclonal antibody and chemotherapy

INTERVENTIONS:
Radiation: neoadjuvant SBRT combined with PD-1 monoclonal antibody and chemotherapy — Eligible participants will receive neoadjuvant treatment consisting of:
  SBRT: One session of 10Gy radiation to the primary tumor, followed by a 150mg subcutaneous injection of pembrolizumab (PD-1 inhibitor).
  Chemotherapy and Immunotherapy: One week after SBRT, participants will undergo 6 cycles of pembrolizumab (400mg), albumin-bound paclitaxel (250mg/m²), and carboplatin (AUC=5).
  Surgery: Surgery will be performed 21 days after the last chemotherapy cycle, with either breast-conserving surgery or modified radical mastectomy. Pathological evaluation will assess the treatment response.
  Adjuvant Immunotherapy: Four weeks post-surgery, patients will receive pembrolizumab every 3 weeks for up to 1 year.
  Other Names: radiotherapy combined with chemotherapy and immunotherapy

SUMMARY:
The primary aim is to evaluate the efficacy of neoadjuvant SBRT combined with PD-1 monoclonal antibody and chemotherapy in patients with triple-negative breast cancer, with the endpoint being the pCR rate-defined as the proportion of patients with no residual invasive cancer in the breast and no axillary lymph node metastasis after treatment. This is a single-arm study. Eligible participants will receive : neoadjuvant treatment consisting of SBRT followed by Envafolimab (PD-1 inhibitor), chemotherapy and immunotherapy (Envafolimab). Surgery will be performed after the last chemotherapy cycle. Pathological evaluation will assess the treatment response. Patients will receive adjuvant immunotherapy (Envafolimab) up to 1 year post-surgery.

ELIGIBILITY:
Inclusion Criteria

Signed written informed consent prior to enrollment

Age ≥ 18 years

ECOG PS score 0-1

Newly diagnosed T1c N1-2 or T2-3 N0-2 breast cancer

Triple-negative breast cancer with PD-L1 CPS < 10

Hemoglobin ≥ 10.0 g/dl, neutrophils ≥ 1.5 × 10⁹/L, platelet count ≥ 100 × 10⁹/L

BUN ≤ 1.5 × upper limit of normal (ULN), creatinine ≤ 1.5 × ULN

Serum bilirubin ≤ 1.5 × ULN, alkaline phosphatase (AKP), AST, and ALT ≤ 2.5 × ULN

Women of childbearing potential must be willing to use contraception during the study

Negative serum or urine pregnancy test within 7 days prior to treatment

Exclusion Criteria

Occult breast cancer

Bilateral breast cancer

Breast tumor unsuitable for SBRT

Unable to undergo MRI scanning

History of other malignancies that may affect survival

Active autoimmune disease or history of autoimmune disease

Current use of immunosuppressants or systemic steroids (within 2 weeks prior to enrollment)

Known allergy to any component of the investigational drugs

Uncontrolled cardiac symptoms or diseases

Active infection or unexplained fever > 38.5°C during screening/before first dose

Other factors likely to cause early study termination (e.g., serious concurrent illnesses, significant lab abnormalities, or social/family circumstances affecting safety/data collection)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
the efficacy of neoadjuvant SBRT combined with PD-1 monoclonal antibody and chemotherapy | From enrollment to the completion of surgery
  pCR rate-defined as the proportion of patients with no residual invasive cancer in the breast and no axillary lymph node metastasis after treatment

IPD SHARING:
Plan to Share IPD: No